CLINICAL TRIAL: NCT05039359
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial of Flecainide Acetate Inhalation Solution for Cardioversion of Recent-Onset, Symptomatic Atrial Fibrillation to Sinus Rhythm
Brief Title: Flecainide Acetate Inhalation Solution for Cardioversion of Recent-Onset, Symptomatic Atrial Fibrillation
Acronym: RESTORE-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Limited efficacy upon blinded review
Sponsor: InCarda Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLE-007
Record Dates: First submitted 2021-08-09; First posted 2021-09-09 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FlecIH-103 (flecainide acetate inhalation solution) (Active Comparator): Up to two 3.5-minute inhalations separated by a 1-minute break, for a total duration of up to 8 minutes on Day 1. Dosing will continue until conversion of AF to SR is observed for ≥1 minute or the full dose (120 mg eTLD) is administered, whichever occurs first.
  Interventions: Drug: FlecIH-103
- Vehicle-matched inhalation solution (placebo) (Placebo Comparator): Up to two 3.5-minute inhalations separated by a 1-minute break, for a total duration of up to 8 minutes on Day 1.
  Interventions: Drug: FlecIH-103

INTERVENTIONS:
Drug: FlecIH-103 — flecainide acetate inhalation solution

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled clinical study designed to evaluate the efficacy and safety of FlecIH-103 (flecainide acetate inhalation solution) compared with placebo in patients with recent-onset, symptomatic newly diagnosed or paroxysmal AF. Approximately 400 patients are expected to be enrolled in this study. Patients will be randomized 3:1 to receive FlecIH-103 at a total dose of up to 120 mg estimated total lung dose (eTLD) (n=300) or placebo inhalation solution (n=100). Randomization will be stratified by geographic region (US and ex-US) and duration of symptoms of the current AF episode (≥1 hour to ≤24 hours and >24 hours to ≤48 hours).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled clinical study designed to evaluate the efficacy and safety of FlecIH-103 (flecainide acetate inhalation solution) compared with placebo in patients with recent-onset, symptomatic newly diagnosed or paroxysmal AF. Approximately 400 patients are expected to be enrolled in this study. The study will consist of the following periods: Screening, Observation, and Follow-up.

The Screening Period comprises the time from the patient signing informed consent to the time of randomization. Screening begins at least 45 minutes prior to dosing and may be extended as needed due to site logistics. During screening, the patient will be evaluated for study eligibility, have a standard triplicate 12-lead ECG to confirm the diagnosis of AF, have a single-lead patch electrode applied for continuous ECG (cECG) recording, undergo a targeted physical examination (including cardiovascular and respiratory systems), have blood drawn for laboratory assessments and a predose pharmacokinetic (PK) sample, have their AF-related symptoms assessed, have vital signs assessed periodically, and be monitored via telemetry to ensure they remain predominantly in AF prior to dosing (ie, no period of SR ≥1 minute in duration or any abnormal rhythm other than AF). After confirmation that the patient meets all applicable eligibility criteria, randomization will take place using a central randomization system. The patient is considered enrolled at the time of randomization.

The Observation Period comprises the time from randomization through 90 minutes after initiation of dosing. After randomization and just prior to the start of dosing (T0), the patient's AF will again be confirmed by a standard triplicate 12-lead ECG; patients who are not in AF at this time must be withdrawn. The patient will inhale the study drug until conversion of AF to SR occurs for ≥1 minute or the complete dose is administered, whichever occurs first. The complete dose of study drug comprises 2 separate 3.5-minute inhalations separated by a 1-minute break. Telemetric recording of ECG and cECG monitoring will continue and vital signs will be monitored periodically. A PK sample will be collected 2 minutes after completion of dosing followed by another standard triplicate ECG collected 5 minutes after completion of dosing. Finally, AF-related symptoms will be checked and a final PK sample will be collected at 90 minutes after initiation of dosing. Wherever a time point requires collection of ECG and/or vital signs in addition to a PK sample, the PK sample is collected last.

If the patient's AF converts to SR (sustained for ≥1 minute) as observed on telemetry during the Observation Period, vital signs and a standard triplicate 12-lead ECG will be recorded immediately following the time of conversion. The Investigator may not offer the patient another rhythm control therapy to cardiovert their AF to SR until after 90 minutes after initiation of dosing. At the end of the Observation Period (ie, 90 minutes after initiation of dosing), the cECG patch will be removed and a standard triplicate 12 lead ECG will be recorded. If the patient's AF converts to SR (sustained for ≥1 minute) after the Observation Period but prior to discharge (eg, due to ECV or other PCV), a standard triplicate 12-lead ECG will be recorded at the time of conversion.

The patient may be discharged per the Investigator's discretion any time after completion of the 90-minute time point assessments. If patient discharge occurs >1 hour after completion of the last 90-minute time point assessment, all 90-minute time point assessments must be repeated just prior to discharge, excluding the PK sample.

The Follow-Up Period consists of 2 follow-up telephone contacts: one at 24 (+12) hours after initiation of dosing, and one at 96 (±24) hours after initiation of dosing. The patient will also be given contact information and be instructed to contact the clinic in the event that any AF-related symptoms occur before these scheduled contact times. Follow-up contacts may also be performed by video call or in-person if the patient is at the clinic. During each follow-up contact, the patient will be queried for concomitant medications and procedures, AEs, AF-related symptoms, and AF-related interventions. End of study coincides with the 96-hour follow-up contact.

An independent Data Monitoring Committee (DMC) will monitor safety throughout the study. An independent Clinical Events Committee (CEC) will review blinded data to adjudicate the primary and several secondary efficacy endpoints and to adjudicate CV events of special interest (ie, hypotension, ventricular tachycardia, bradycardia, sinus pause, atrial flutter with 1:1 conduction, and other arrhythmias).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤85 years of age
2. Recent onset of symptomatic newly diagnosed or paroxysmal AF

   1. Recent onset is defined as a symptom duration ≥1 and ≤48 hours at time of dosing
   2. Newly diagnosed AF is AF that has not been diagnosed previously, independent of its duration
   3. Paroxysmal AF is defined as recurrent AF in a patient whose previous AF episode(s) self-terminated (ie, without treatment) or terminated with intervention ≤7 days of onset.
   4. A symptomatic recent-onset AF episode post cardiac ablation for paroxysmal AF would be considered eligible

Exclusion Criteria:

1. History of non self-terminating AF/AFL as defined by

   1. One or more failed attempts to restore SR with pharmacological therapy
   2. ECV procedure for an AF episode ≤1 year prior to screening. Exception: One (1) prior ECV is allowed if no option for pharmacological conversion was previously available
   3. More than 3 ECV procedures in ≤5 years prior to screening
2. Current diagnosis of persistent AF

   1. Persistent AF defined as AF that is continuously sustained >7 days, including episodes terminated by cardioversion (drugs or electrical cardioversion) after >7 days. Patients with persistent AF do not have self-terminating AF episodes
   2. Patients who have undergone an ablation procedure for persistent AF are not eligible
3. One or more episodes of AFL ≤6 months prior to randomization

   a. Exception: a patient who has received ablation for AFL ≤3 months prior to screening with no recurrence of AFL prior to randomization is considered eligible Vital signs
4. Hemodynamic or cardiac instability during AF, defined as any of the following:

   1. Systolic blood pressure <100 or ≥160 mmHg
   2. Diastolic blood pressure ≥95 mmHg
   3. Ventricular heart rate <80 or >160 bpm
5. Respiratory rate >22 breaths per minute Relevant structural heart disease
6. History of decompensated heart failure (HF)
7. Evidence of significant HF defined as any of the following:

   a. Hospitalization in the last 12 months for HF or suspected HF event b. Most recent assessment of left ventricular ejection fraction (LVEF) <45% i. For patients in the United States, a standard diagnostic echocardiogram assessed ≤180 days prior to screening is required to ascertain eligibility. If none is available, the patient must undergo a standard diagnostic echocardiogram or a diagnostic echocardiogram using a portable ultrasound device (handheld echocardiogram [HHE]) during screening to confirm eligibility c. New York Heart Association (NYHA) Class II-IV symptoms d. Medication history suggestive of HF per the Investigator's discretion
8. Signs or symptoms of ongoing myocardial ischemia, including any of the following:

   1. Significant ST segment elevation or depression (ie, ≥2 mm) on a standard 12-lead ECG
   2. Echocardiogram findings (eg, wall motion abnormalities) suggestive of acute myocardial infarction (MI)
   3. Angina pectoris, atypical angina pectoris, or receiving antianginal medication for ischemia
9. History of MI ≤3 months of screening
10. History of uncorrected moderate or severe aortic or mitral valvular stenosis, in the opinion of the Investigator

    a. If an echocardiogram is performed at screening, moderate or severe valve disease observed during the examination is considered exclusionary
11. History of LV hypertrophy with LV thickness >12 mm as observed in the most recent assessment, ie, an echocardiogram Other CV conditions
12. Stroke (including transient ischemic attack) ≤3 months prior to randomization
13. History of any of the following cardiac abnormalities:

    1. Long QT syndrome
    2. Conduction system disease (eg, PR interval >200 ms, second- or third degree heart block, bundle branch block)
    3. Brugada syndrome
    4. Torsade de pointes
    5. Diagnosed with sinus node dysfunction (eg, sick sinus syndrome) or any of the following:

    i. History of unexplained or cardiovascular syncope ii. Bradycardia suggestive of sinus node dysfunction iii. Prior electrical or pharmacological cardioversion associated with sinus or ventricular pause >3 seconds or ventricular heart rate <45 bpm at time of conversion
14. Any of the following ECG-related features at screening:

    1. QT interval corrected for heart rate using the Fridericia formula (QTcF) >480 msec
    2. Wide QRS complex (ie, duration ≥120 msec) or history of documented wide QRS complex tachycardia (ie, wide QRS complex with ventricular heart rate >100 bpm)
    3. Presence of ventricular tachycardia (VT). Site telemetry should be equipped with an alarm system for VT and PVCs or be continuously visually observed prior to dosing
15. Presence of a pacemaker
16. Cardiac surgery for any of the exclusionary conditions (eg, valvular disease, hypertrophy, coronary artery disease) ≤6 months prior to randomization Prior and concomitant non-CV conditions
17. Known severe renal impairment or patient receiving dialysis
18. Known abnormal liver function, including hepatic disease or biochemical evidence of significant liver derangement
19. Uncorrected hypokalemia

    1. Hypokalemia is defined as serum potassium below the normal range according to the local laboratory reference ranges at screening
    2. If serum potassium is below the normal range at screening, therapeutic correction (eg, potassium supplementation) is required
20. Uncorrected hypomagnesemia

    1. Hypomagnesemia is defined as serum magnesium below the normal range according to the local laboratory reference ranges at screening
    2. If serum magnesium result is below the normal range at screening, therapeutic correction (eg, magnesium supplementation) is required
21. Chronic obstructive pulmonary disease or other established pulmonary disease in need of inhalation medication

    a. Exception: patients with intermittent mild asthma who are not experiencing active symptoms at screening, and whose asthma is well controlled with as-needed administration of a bronchodilator ≤2 days/week, and who has not experienced ≥2 exacerbations requiring oral systemic corticosteroids ≤1 year prior to screening
22. History of bronchospasm (eg, hyperreactive airways to inhalants) or difficulty inhaling medications
23. Previous or current hospitalization for COVID-19, or any secondary cardiomyopathy from COVID-19 Prior and concomitant medications and procedures
24. Treatment with Class I or III AADs ≤7 days prior to randomization
25. Treatment with amiodarone ≤12 weeks prior to randomization
26. Known hypersensitivity to flecainide acetate, any active metabolites of flecainide acetate, or any excipients in FlecIH-103
27. Any condition or circumstance which in the opinion of the Investigator may make the patient unsuitable for the study, such as:

    1. High risk for stroke based on the screening coagulation panel or medical history per Investigator's discretion (eg, CHA2DS2-VASc score)
    2. Congenital heart disease
    3. AF that is secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause
    4. A serious or life-threatening medical condition
    5. An acute infection
28. Known drug or alcohol dependence ≤12 months prior to screening as judged by the Investigator
29. A body mass index ≥35 kg/m2
30. Legally incompetent to provide informed consent
31. Previous treatment with any other investigational drug ≤30 days from screening or 5 half-lives of the drug, whichever is longer
32. Female of childbearing potential defined as any of the following:

    1. Not surgically sterile or postmenopausal (Appendix 1)
    2. A negative pregnancy test is unavailable at screening
    3. Pregnant or breastfeeding at screening
33. Males whose sexual partners are women of childbearing potential (WOCBP) must use at least one highly effective method of contraception during the study unless permenantly sterile by bilateral orchiectomy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Assessment of proportion of patients whose AF converts using continuous ECG monitoring | 90 minutes
  To compare the efficacy of flecainide acetate inhalation solution and placebo for the conversion of atrial fibrillation (AF) to sinus rhythm (SR) in patients with recent-onset, symptomatic newly diagnosed or paroxysmal AF. Conversion from AF to SR will be monitored via continuous ECG recording. The efficacy of flecainide acetate solution and placebo will be compared using conversion as recorded on the ECG.

SECONDARY OUTCOMES:
Time of conversion to be monitored using continuous ECGs | 90 minutes
  To compare the effects of flecainide acetate inhalation solution and placebo on the time to conversion of AF to SR. Conversion from AF to SR will be monitored via continuous ECG recording. The time of conversion as captured on the continuous ECG will be compared between flecainide acetate inhalation solution and placebo.
Assessing and comparing the AF related symptoms by using a questionnaire | 90 minutes post dose
  To compare the effects of flecainide acetate inhalation solution and placebo on the AF-related symptoms. The AF-related symptoms will be reported by the patients in the AF-Related Symptoms Questionnaire at 90 minutes after initiation of dosing.
Assessing and comparing the hospital admissions between the active vs. placebo | 90 minutes
  To compare the effects of flecainide acetate inhalation solution and placebo on the patient hospitalizations prior to discharge as reported by the investigator in the CRF.
Assessing and comparing the AF-related interventions prior to discharge between the active vs. placebo | 90 minutes
  To compare the effects of flecainide acetate inhalation solution and placebo on the AF-related interventions as reported by the investigator in the CRF.
Assessing and comparing the time of discharge | 90 minutes
  To compare the effects of flecainide acetate inhalation solution and placebo on the time to discharge as reported by the investigator in the CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Belardinelli, MD, Study Director — InCarda Therapeutics, Inc.
Locations (40):
- United States (18):
  - UC Davis Medical Center, Davis, California
  - Memorial Care, Long Beach, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Orlando Health Heart and Vascular Institute and Orlando Regional medical Center, Orlando, Florida
  - Tampa General Hospital; Center of Research Excellence, Tampa, Florida
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - North Kansas City Hospital, Kansas City, Kansas
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Saint Michaels Medical Center, Newark, New Jersey
  - The Valley Hospital, Inc, Ridgewood, New Jersey
  - Mount Sinal Hospital, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Cleveland Clinic Emergency Department, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania
- Czechia (2):
  - EDUMED s.r.o., Náchod
  - Nemocnice Slany, Slaný
- Hungary (2):
  - DPC Hospital Egyesitett Szent Istvan es Szent Laszlo Korhaz, Budapest
  - University of PACs, Pécs
- Netherlands (8):
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Spaarne Gasthuis, Haarlem
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Diakonessenhuis, Utrecht
  - Maxima Medisch Centrum, Veldhoven
- Poland (2):
  - Mazowiecki Szpital Specjalistyczny w Ostrolece, Ostrołęka
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
- Spain (8):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - La Paz Univerisity Hospital, Madrid
  - Hospital Universitario Puera de Hierro, Madrid
  - Fundacion Hospital Son Liatzer, Palma de Mallorca
  - Hospital Santiago De Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rienstra M, Woite-Silva AC, Kuijper A, Eijsbouts S, Kraaier K, Janota T, Van Ofwegen C, Tuininga Y, Badings E, Merino JL, Ruskin JN, Camm AJ, Kowey PR, Dufton C, Maupas J, Parsell D, Belardinelli L. Flecainide acetate inhalation solution for cardioversion of recent-onset, symptomatic atrial fibrillation: results of the phase 3 RESTORE-1 trial. Europace. 2025 Mar 28;27(4):euaf064. doi: 10.1093/europace/euaf064. PMID 40132102